CLINICAL TRIAL: NCT04056299
Title: Phase 2 Study of AR201 Oral Immunotherapy for Desensitization in Children, Adolescents, and Young Adults With Hen Egg Allergy
Brief Title: Oral Immunotherapy for Desensitization in Children, Adolescents, and Young Adults With Hen Egg Allergy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated by the Sponsor based on difficulties in meeting enrollment goals, especially during the COVID-19 pandemic, and not for reasons relating to any concerns regarding quality, safety, or efficacy.
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIME01
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Hen Egg Allergy
Keywords: CODIT™ (characterized oral desensitization immunotherapy™); Hen Egg Allergic Children; Desensitization; AR201; Allergy; Hen Egg Allergy; Characterized Hen Egg Allergen; Oral Immunotherapy; CHEA (Characterized Hen Egg Allergen); Food Allergy
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: 2:1 randomization
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AR201 powder (Active Comparator): Subjects were randomized to active arm of AIME01 and administered AR201 in escalating doses for approximately 6 months, followed by a maintenance dose for approximately 12 weeks
  Interventions: Biological: AR201 powder
- Placebo powder (Placebo Comparator): Subjects were randomized to placebo arm of AIME01 and administered placebo for approximately 6 months, followed by maintenance placebo for approximately 12 weeks.
  Interventions: Biological: Placebo powder

INTERVENTIONS:
Biological: AR201 powder — AR201 powder (Hen Egg allergen formulation) provided in capsules
  Arms: AR201 powder
Biological: Placebo powder — Placebo powder provided in capsules
  Arms: Placebo powder

SUMMARY:
To determine the efficacy and safety of AR201 in a characterized oral desensitization immunotherapy (CODIT™) regimen in hen egg-allergic subjects aged 4 to 26 years, inclusive.

DETAILED DESCRIPTION:
This is a phase 2, randomized, double-blind, placebo-controlled study of the efficacy and safety of AR201 in a CODIT regimen in hen egg-allergic subjects aged 4 to 26 years, inclusive. The study was conducted at 8 sites in the United States.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 4 to 26 years, inclusive
* Written informed consent from subjects, as appropriate per local requirements, and parent/guardian
* Written assent from subjects who are minors, as appropriate per local requirements
* History of physician-diagnosed hen egg allergy
* Elevated egg specific IgE and/or mean wheal diameter on SPT to egg
* Experience dose-limiting symptoms at or before the 300 mg challenge dose of dried egg white protein on Screening DBPCFC
* Use of effective birth control by sexually active female subjects of childbearing potential

Key Exclusion Criteria:

* History of severe or life-threatening anaphylaxis within 60 days before screening
* History of non-IgE mediated hen egg allergy such as food protein-induced enterocolitis syndrome (FPIES)
* History of eosinophilic esophagitis (EoE), other eosinophilic gastrointestinal disease, chronic, recurrent, or severe gastroesophageal reflux disease (GERD), symptoms of dysphagia or recurrent gastrointestinal symptoms of unknown etiology
* History of a mast cell disorder including systemic mastocytosis, urticaria pigmentosa, chronic idiopathic or chronic physical urticaria beyond simple dermatographism (e.g., cold urticaria, cholinergic urticaria), and hereditary or idiopathic angioedema
* History of chronic disease (except asthma, atopic dermatitis, or allergic rhinitis) which may require a change in immunosuppressive medication regimen or chronic corticosteroid use
* History of cardiovascular disease, including uncontrolled or inadequately controlled hypertension
* Developing dose-limiting symptoms to placebo challenge during the Screening DBPCFC
* Having the same place of residence as another subject in the study
* Any other condition that, in the opinion of the Investigator, precludes participation for reasons of safety

Ages: 4 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director of Regulatory Affairs, Study Chair — Aimmune Therapeutics, Inc.
Locations (11):
- United States (11):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Allergy & Asthma Medical Group and Research Center, A.P.C, San Diego, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - Allergy and Asthma Clinical Research dba Bay Area Allergy, Walnut Creek, California
  - Atlanta Allergy & Asthma Clinic, PA, Marietta, Georgia
  - Idaho Allergy LLC, dba Idaho Allergy and Research, Eagle, Idaho
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - Clinical Research Institute Inc, Minneapolis, Minnesota
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Seattle Allergy & Asthma Research Institute dba ASTHMA, Inc. Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AR201 Powder | Placebo Powder
Started | 9 | 6
Completed | 6 | 3
Not Completed | 3 | 3
Not completed — Sponsor discontinued study | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AR201 Powder | Placebo Powder | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Median (Full Range); unit: years] | 13.0 [6 to 23] | 5.5 [4 to 12] | 7.0 [4 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Tolerating a Single Highest Dose of at Least 1000 mg Dried Egg White Protein With no More Than Mild Symptoms at the Exit Double-blind Placebo Controlled Food Challenge (DBPCFC)
Time Frame: 9-12 months
Population: The study was prematurely terminated due to difficulties in meeting enrollment goals due to the Coronavirus Disease 2019 (COVID-19) pandemic. As a consequence, all prespecified efficacy endpoint analysis were not performed, and the exit DBPCFC was optional and limited to subjects who completed at least 9 months of study treatment including at least 4 weeks at 300 mg/day, and tolerated the 300 mg/day dose for approximately 2 consecutive weeks before the exit DBPCFC.
Measure: Count of Participants; unit: Participants
Groups:
- AR201 Powder: Study product provided as dried egg white in pull-apart capsules.
  AR201 powder in capsules: AR201 powder (Hen Egg allergen formulation) formulated to contain dried egg white at different dosage strengths.
- Placebo Powder: Placebo formulation in pull-apart capsules containing only inactive ingredients
  Placebo powder provided in capsules: Placebo powder formulated to match the color and texture of dried egg white.
Arm/Group | AR201 Powder | Placebo Powder
Number analyzed (Participants) | 9 | 6
Participants | 1 | 0

2. Secondary Outcome: Number of Participants by Maximum Dose Achieved With no or Mild Symptoms at Exit DBPCFC
Time Frame: 9-12 months
Population: The study was prematurely terminated due to difficulties in meeting enrollment goals due to the COVID-19 pandemic. As a consequence, all prespecified efficacy endpoint analysis were not performed, and the exit DBPCFC was optional and limited to subjects who completed at least 9 months of study treatment including at least 4 weeks at 300 mg/day, and tolerated the 300 mg/day dose for approximately 2 consecutive weeks before the exit DBPCFC.
Measure: Count of Participants; unit: Participants
Arm/Group | AR201 Powder | Placebo Powder
Number analyzed (Participants) | 9 | 6
Participants
  None | 0 | 0
  1 mg | 0 | 0
  3 mg | 0 | 0
  10 mg | 0 | 0
  30 mg | 0 | 0
  100 mg | 0 | 0
  300 mg | 2 | 0
  600 mg | 0 | 0
  1000 mg | 0 | 0
  2000 mg | 1 | 0
  Did not have an exit DBPCFC | 6 | 6

ADVERSE EVENTS:
Time Frame: Approximately 9 months
Arm/Group | AR201 Powder | Placebo Powder
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/6
Other Adverse Events (participants affected / at risk) | 9/9 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR201 Powder (N=9) | Placebo Powder (N=6)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR201 Powder (N=9) | Placebo Powder (N=6)
Abdominal pain (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Lip pruritus (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Oral pruritus (Gastrointestinal disorders) | 1 | 2
Tongue pruritus (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 1
Blepharitis (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1
Merycism (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (1):
  • Study Protocol (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT04056299/Prot_000.pdf